CLINICAL TRIAL: NCT04666636
Title: Mechanisms for Activation of Beige Adipose Tissue in Humans
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Philip Kern (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Philip Kern, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 60821; R01DK124626 (NIH)
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-10

CONDITIONS: PreDiabetes
Keywords: beige; adipose; glucose; fat; BAT; diabetes; metabolism; DEXA
MeSH Terms: conditions — Prediabetic State; Platelet Glycoprotein IV Deficiency; Diabetes Mellitus | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants in the group will receive placebo.
  Interventions: Drug: Placebo
- Mirabegron (Experimental): Participants in this group will receive Mirabegron for 16 weeks.
  Interventions: Drug: Mirabegron
- Sub-Study: Mirabegron and the acute response to food (Experimental): This sub-study will involve the recruiting of the same subjects who are eligible for this study as described above. Subjects will report to the CCTS fasting on 3 separate days. On each visit, the subject will have 5 blood draws and each blood draw will be about 8 ml, for a total of 40 ml of blood at each visit. Visit 1 will involve the participant consuming a standardized meal. At visit 2, participants will take 50mg of Mirabegron. And visit 3 will involve the participant consuming the same meal as visit 1 and also taking 50 mg of mirabegron.
  Interventions: Drug: Mirabegron 50 MG
- Sub-Study: Mirabegron dosing and Oral Glucose Tolerance Tests (Optional) (Experimental): Studies have found that larger doses of mirabegron do not elicit the same improvements in insulin sensitivity. Therefore, we aim to perform a dose-response study to gain an improved understanding of mirabegron dosing and changes in insulin sensitivity.
  This sub-study will have 4 total visits. visit 1 is a baseline oral glucose tolerance test. At the end of visit 1, participants will be given 6 weeks of mirabegron (25 mg) and will take 1 pill once per day for 4-6 weeks leading up to visit 2. Visit 2 will also be a standard oral glucose tolerance test. At the end of visit 2, participants will be given 6 weeks of mirabegron (50 mg) and take 1 pill once per day for 4-6 weeks leading up to visit 3. Visit 3 will also be a standard oral glucose tolerance test. At the end of visit 3, participants will be given 6 weeks of mirabegron (10 mg) and take 1 pill once per day for 4-6 weeks. Visit 4 will be the final visit and will also be a standard oral glucose tolerance test.
  Interventions: Drug: Mirabegron 100 mg

INTERVENTIONS:
Drug: Placebo — Participants will take one pill (placebo) daily for the first week and two pills daily for the remaining 15 weeks.
  Arms: Placebo
Drug: Mirabegron — Participants will take one pill (50mg Mirabegron) daily for the first week. For week two, participants will take two pills (50mg and 25mg Mirabegron). Unless there are side effects, for the remaining 14 weeks participants will take two pills (50mg each) daily.
  Other Names: Myrbetriq
  Arms: Mirabegron
Drug: Mirabegron 50 MG — Participants will take one pill (50mg Mirabegron) daily between visit 2 and visit 3
  Other Names: Myrbetriq
  Arms: Sub-Study: Mirabegron and the acute response to food
Drug: Mirabegron 100 mg — participants will be given 6 weeks of mirabegron (25 mg) and will take 1 pill once per day for 4-6 weeks. Next participants will be given 6 weeks of mirabegron (50 mg) and take 1 pill once per day for 4-6 weeks. Last participants will be given 6 weeks of mirabegron (100 mg) and take 1 pill once per day for 4-6 weeks.
  Other Names: Myrbetriq
  Arms: Sub-Study: Mirabegron dosing and Oral Glucose Tolerance Tests (Optional)

SUMMARY:
Mirabegron (Myrbetriq®, Astellas) is a highly specific and well-tolerated ß3 agonist marketed for overactive bladder. This trial will assess the effects of mirabegron on glucose tolerance and adipose tissue in prediabetic patients

DETAILED DESCRIPTION:
Among the many survival adaptations developed by mammals is a defense against the cold and hypothermia; one of these adaptations is the ability to uncouple oxidative phosphorylation and generate heat, rather than adenosine triphosphate (ATP), from lipid substrate in specialized tissues, and there has been much interest in exploiting this inefficient metabolism for the treatment of obesity and insulin resistance. Brown adipose tissue (BAT) protects against obesity in mice, and studies have documented cold-induced BAT in humans using positron emission tomography (PET-CT) scanning. Additional studies have demonstrated that white adipose tissue (WAT) can upregulate its thermogenic capacity and become "beige", and this beiging of SC WAT likely provides an additional defense against the cold.

Brown and beige fat can be activated by cold temperatures, or through catecholamines. The catecholamines epinephrine and norepinephrine have undesirable side effects. However, adipocytes are among the few cells that contain ß3 adrenergic receptors (ß3AR), whereas the heart is dominated by ß1 and ß2 receptors. Therefore, a drug that could target the ß3AR could activate brown/beige fat without cardiovascular side effects. Recently, there have been human studies performed and obese human subjects participants were treated with the ß3AR agonist mirabegron. This resulted in improved glucose homeostasis by increasing insulin sensitivity and insulin secretion. It was also found that mirabegron treatment of obese adults did not increase BAT or induce weight loss, but instead induced beige fat, along with increased insulin sensitivity, which was accompanied by an increase in type I fibers in skeletal muscle. Mirabegron treatment stimulated subcutaneous (SC) WAT beiging, lipolysis, and remodeling. However, unlike WAT, insulin-producing ß-cells and muscle do not express the ß3AR; therefore, it is thought that the beneficial effects of mirabegron treatment occurred by an indirect mechanism.

Currently, mirabegron (Myrbetriq®, Astellas) is a highly specific and well-tolerated ß3 agonist marketed for overactive bladder. It is hypothesized that mirabegron treatment of prediabetic subjects will improve glucose homeostasis through improved insulin sensitivity and ß-cell function, in addition to other changes in adipose tissue. Additionally, mirabegron treatment may change the plasma composition of proteins, lipids, metabolites, short-chain fatty acids, or exosomal miRNAs that are known to affect peripheral tissue function.

This trial will quantify the effects of the ß3 agonist mirabegron on glucose metabolism and adipose tissue in a placebo-controlled trial and determine some of the mechanistic underpinnings of these effects.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-45
* prediabetes (A1c 5.7-6.4)
* impaired fasting glucose or impaired glucose tolerance

Exclusion Criteria:

* diabetes
* chronic use of anti-diabetic medication
* acute or chronic inflammatory condition
* unstable medical condition
* cancer
* renal insufficiency
* any contraindication for Mirabegron
* BMI >45

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Glucose Tolerance | 16 weeks (at baseline and at 16 weeks)
  The standard oral glucose tolerance test (OGTT) using 75g glucose will be used to assess tolerance.
Change in Body Composition | 16 weeks (at baseline and at 16 weeks)
  Body composition (percent body fat) will be measured using dual-energy X-ray absorptiometry (DEXA).
Change in Resting Metabolic Rate | 16 weeks (at baseline and at 16 weeks)
  Resting Metabolic Rate (RMR) will be measured using indirect calorimetry.
Change in Brown Adipose Tissue Activity | 16 weeks (at baseline and at 16 weeks)
  Brown adipose tissue (BAT) activity will be measured using water-vest cold stimulation combined with positron emission tomography (PET-CT).
Change in Peripheral Insulin Sensitivity | 16 weeks (at baseline and at 16 weeks)
  Peripheral insulin sensitivity will be measured with a euglycemic clamp.
Change in Insulin Secretion | 16 weeks (at baseline and at 16 weeks)
  Insulin secretion will be measured with a euglycemic clamp.
Change in glycohemoglobin | 16 weeks (at baseline and at 16 weeks)
  Hemoglobin A1c (HbA1C) will be measured from blood samples.
Change in Matsuda Index for Dosing Sub Study | Baseline, week 6, week 12, week 18
  Comparison of change in Matsuda Index as determined by 2-h oral glucose tolerance test (OGTT). During OGTT, response to oral 75g glucose intake is determined by measuring insulin and glucose in timed samples obtained at 0, 30, 60, 90 and 120 min. Increase in scores reflect improvement in whole body insulin sensitivity.
Change in bile acids/blood proteins | Baseline, week 1, week 2
  FGF-19 and total bile acids will be analyzed and compared across the different conditions. Plasma bile acid concentration (ng/mL) will be measured and compared across the different doses of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kern, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No